CLINICAL TRIAL: NCT06168461
Title: Aspirin for the Treatment of Vascular Dysfunction After Preeclampsia
Brief Title: Daily Aspirin Treatment After Preeclampsia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anna Stanhewicz, PhD (Other)
Responsible Party: Sponsor-Investigator, Anna Stanhewicz, PhD, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 202303799
Record Dates: First submitted 2023-09-13; First posted 2023-12-13 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Preeclampsia
Keywords: preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): placebo pill taken once daily at bedtime for 12 weeks
  Interventions: Drug: Placebo
- aspirin (Experimental): 162mg aspirin taken once daily at bedtime for 12 weeks
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — 162mg aspirin capsule
  Arms: aspirin
Drug: Placebo — placebo capsule
  Arms: placebo

SUMMARY:
Women who develop preeclampsia during pregnancy are four times more likely to develop cardiovascular disease later in life, even if they are otherwise healthy. The reason why this occurs may be related to lasting blood vessel damage after the pregnancy but there are currently no specific treatment strategies to prevent this disease progression. This study addresses this public health issue by examining whether starting low dose aspirin therapy after pregnancy is an effective treatment for lasting blood vessel damage in order to inform better clinical management of cardiovascular disease risk in women who have had preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* had preeclampsia in the past 5 years,
* 18 years or older

Exclusion criteria:

* current daily aspirin use,
* skin diseases,
* current tobacco or nicotine use (including vaping),
* diagnosed or suspected hepatic or metabolic disease including chronic kidney disease (CKD) defined as reduced eGFR < 60 mL/min/1.73m2,
* statin or other cholesterol-lowering medication,
* current antihypertensive medication,
* history of hypertension prior to pregnancy,
* history of gestational diabetes,
* currently pregnancy,
* body mass index <18.5 kg/m2,
* allergy to materials used during the experiment.(e.g. latex),
* known allergies to study drugs,
* bleeding disorders, peptic ulcer disease, gastritis, GI bleeding and gastroesophageal reflux disease (GERD).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
magnitude of microvascular endothelial function | baseline, 12 weeks
  skin blood flow response to acetylcholine delivered via intradermal microdialysis
magnitude of brachial artery endothelial function | baseline, 12 weeks
  brachial artery flow mediated dilation
magnitude of microvascular endothelin-1 mediated constriction | baseline, 12 weeks
  skin blood flow response to endothelin-1 delivered via intradermal microdialysis

SECONDARY OUTCOMES:
magnitude of microvascular nitric oxide-dependent dilation | baseline, 12 weeks
  skin blood flow response to acetylcholine + L-NAME delivered via intradermal microdialysis

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States